CLINICAL TRIAL: NCT07286318
Title: A Randomized Controlled Trial of Topical 5% Niacinamide for Skin Cancer Prevention in Transplant Recipients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Marissa Lobl (Other)
Responsible Party: Sponsor-Investigator, Marissa Lobl, UPMC Dermatology Resident, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY25050043
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Skin Cancer; Cutaneous Squamous Cell Carcinoma (CSCC); Actinic Keratosis (AK); Organ Transplant Recipient
Keywords: Niacinamide; Cutaneous squamous cell carcinoma; Basal cell carcinoma; Organ transplant recipient; Actinic keratosis
MeSH Terms: conditions — Skin Neoplasms; Keratosis, Actinic; Carcinoma, Basal Cell | interventions — Niacinamide; Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sunscreen Only (Active Comparator): The participants will not be assigned to any intervention. They will use broad spectrum SPF 30 daily sunscreen as instructed regardless of whether or not they are enrolled in the study.
  Interventions: Drug: Sunscreen
- Sunscreen + Niacinamide (Experimental): In addition to using broad spectrum SPF 30 daily sunscreens, participants will apply topical 5% niacinamide daily to any sun exposed areas.
  Interventions: Drug: Topical niacinamide 5% cream; Drug: Sunscreen

INTERVENTIONS:
Drug: Topical niacinamide 5% cream — Participants will be instructed to apply topical 5% niacinamide daily to any sun exposed areas.
  Arms: Sunscreen + Niacinamide
Drug: Sunscreen — Sunscreen application daily, broad spectrum SPF 30, to any sun exposed areas

SUMMARY:
A Randomized Controlled Trial of Topical 5% Niacinamide for Skin Cancer Prevention in Organ Transplant Recipients

This study is designed to evaluate whether a topical 5% niacinamide cream can help prevent skin cancer in organ transplant recipients. Individuals who have received an organ transplant have a much higher risk of developing precancerous skin growths and skin cancers because of long-term immune-suppressing medications. Although sunscreen is an important part of sun protection, additional preventive approaches are needed. Early research suggests that niacinamide may help protect the skin, and this trial will examine whether a topical formulation provides benefit in this high-risk group.

The study will test whether daily use of topical 5% niacinamide reduces the number of actinic keratoses over 6 and 12 months and whether it decreases the development of new keratinocyte cancers when compared with sunscreen alone. The study will also evaluate how well the topical product is tolerated and whether it can be used consistently as part of a daily skin-care routine.

A total of 20 adult organ transplant recipients with a history of multiple actinic keratoses and at least one prior non-melanoma skin cancer will enroll in this 12-month, randomized, controlled trial. Participants will be assigned to receive either daily topical 5% niacinamide plus sunscreen or sunscreen alone. Skin examinations will be performed at 6 and 12 months using standardized mapping methods. Information on treatment tolerability, adherence, and any side effects will be collected through structured surveys, and any lesions suspicious for cancer will be evaluated by a board-certified pathologist.

DETAILED DESCRIPTION:
Background, Significance, and Preliminary Studies

Organ transplant recipients (OTRs) have at least a 50 times higher risk of developing non-melanoma skin cancers than the general population (Moloney et al., 2006). These skin cancers in OTRs also tend to be more aggressive, with higher rates of recurrence and metastasis (Martinez et al., 2003). Immunosuppression in OTRs is primarily achieved through the use of pharmacologic agents such as mycophenolate mofetil, azathioprine, cyclosporine, and tacrolimus, among other medications. These agents work by inhibiting various components of the immune system to prevent graft rejection. For instance, calcineurin inhibitors like cyclosporine and tacrolimus inhibit T-cell activation by blocking the production of interleukin-2 (IL-2), a critical cytokine for T-cell proliferation. Mycophenolate mofetil and azathioprine inhibit purine synthesis, thereby reducing lymphocyte proliferation. These immunosuppressive drugs, while effective in preventing rejection, also impair DNA repair mechanisms and immune surveillance and increase the risk of malignancies, particularly skin cancers.

Nicotinamide (NAM), the amide derivative of vitamin B3, has been investigated for its potential role in reducing the incidence of skin cancer. Ultraviolet (UV) radiation exposure in the absence of NAM results in a significant reduction in cellular adenosine triphosphate (ATP) levels. NAM has been shown to enhance DNA repair mechanisms and mitigate UV-induced immunosuppression by preserving cellular ATP levels (Park et al., 2010). In the context of oncogenesis, the maintenance of ATP levels is commonly associated with the promotion of antitumor immune responses, whereas elevated levels of extracellular adenosine (ADO) are often seen in cancer. The ectonucleotidase CD39 catalyzes the rate-limiting step in the hydrolysis of extracellular ATP to extracellular ADO. Work by Whitley et al. (2021), employing a murine model, demonstrated that CD39 expression on skin-resident T cells regulates DNA damage repair through ATP-mediated signaling pathways. Taken together, these findings suggest a mechanistic pathway by which NAM may exert chemopreventive effects. NAM appears to maintain cellular ATP levels, which facilitates DNA repair and supports antitumor immunity through the modulation of extracellular ATP and adenosine (ADO) signaling.

Several other potential mechanisms by which NAM may be chemoprotective are described in the literature. In human keratinocyte cultures, tumor protein p53 (TP53), a key protector of the DNA damage response, was significantly upregulated following UV exposure in the presence of NAM when compared to UV exposure without NAM (Sirapivabu et al., 2009). TP53 is often referred to as the guardian of the genome and its loss is observed in many cancers. Further, keratinocytes treated with NAM and exposed to UV radiation and arsenic demonstrated protection against cyclobutane pyrimidine dimer (CPDs) and 8-oxo-7,8-dihydro-2'-deoxyguanosine formation, which are DNA photolesions (Damian et al., 2015). Photolesions can result in carcinogenic mutations if not repaired. NAM has also been shown to facilitate repair of such photolesions through multiple pathways (Surjana et al., 2013).

While oral NAM has shown promise in skin cancer prevention, clinical trials in high-risk patients have yielded mixed results. A phase 3 randomized controlled trial by Chen et al. (2015) of 386 high-risk immunocompetent patients demonstrated that oral nicotinamide (500 mg twice daily for 12 months) significantly reduced the rate of new nonmelanoma skin cancers (NMSCs) by 23% (P = 0.02) compared to placebo. Reductions were observed for new squamous cell carcinomas (30% reduction, P = 0.05) and basal cell carcinomas (20% reduction, P = 0.12), and actinic keratoses counts were significantly lower throughout treatment (P < 0.001 at multiple time points). A pilot double-blind randomized trial in renal transplant patients by Chen et al. (2016) evaluated oral nicotinamide (500 mg twice daily) for prevention of nonmelanoma skin cancers (NMSCs) and actinic keratoses (AKs). Over 6 months, nicotinamide showed a nonsignificant 35% relative reduction in NMSC rate (P = 0.36) and a 16% reduction in AKs (P = 0.15) compared to placebo. A study by Hwang et al. (2025) utilized a retrospective cohort study design to evaluate the effect of oral nicotinamide supplementation in a group of 47 OTRs. It was demonstrated that nicotinamide 500 mg twice daily for at least a year decreased the incidence of KCs at one and two year follow up (Hwang et al., 2025).

However, the beneficial effects observed in these studies have not been consistent throughout the literature. A recent phase 3 randomized trial by Allen et al. (2023) evaluated oral nicotinamide (vitamin B3) for skin cancer chemoprevention in OTRs. Despite previous promising results in immunocompetent individuals, the study found no significant reduction in new AKs with oral NAM over 12 months compared to placebo (Allen et al., 2023). However, while not statistically significant, a notable trend toward reduced invasive squamous cell carcinoma (SCC) was observed in the NAM treated patients. In addition, this study has significant limitations as it terminated early due to poor recruitment. Another small, randomized trial of 30 patients by Zhang et al. (2023) evaluated oral NAM for preventing AKs in kidney transplant recipients with prior keratinocyte carcinoma. The study found no significant reduction in AK development with oral NAM (500 mg twice daily) over 12 months compared to placebo. Tolerability issues led to dose reduction and higher attrition in the NAM group, highlighting challenges with systemic therapy in this population. These findings underscore the need to investigate alternative and synergistic approaches, such as topical niacinamide, which may improve tolerability and localized efficacy for skin cancer prevention in transplant recipients.

Topical niacinamide offers an exciting alternative and possible adjunct chemopreventive strategy for transplant patients. By directly targeting the skin, sunscreen containing topical niacinamide has been shown to prevent UV-induced immunosuppression by altering multiple pathways similar to the oral form including cell cycle, apoptosis, immunoregulation, and cellular energy (Torres-Moral et al., 2024) Topical niacinamide's excellent safety profile and localized action make it a promising additional or standalone approach for skin cancer chemoprevention in high-risk populations. Further studies would be helpful to explore its full potential in transplant dermatology.

Preliminary studies by our group are evaluating transplant patients' medication preferences and openness to try a product with topical niacinamide to potentially decrease risk for skin cancer. A pilot dataset from our group (n=10) demonstrated that oral medication use is high, with 8/10 participants taking seven or more medications daily. Concerns about oral medications are notable, with 7/10 participants reported being concerned or somewhat concerned about side effects, and 6/10 being concerned or somewhat concerned with drug interactions. Use of topical medications is less prevalent, with 8/10 participants using 0-1 per day and there were fewer concerns with interactions and side effects. When informed about the potential skin cancer prevention benefits of topical niacinamide, 7/10 participants reported that they would be very or somewhat likely to try this in their daily routine. The key factor influencing willingness to try such a product was recommendation from a healthcare provider, selected by 9/10 patients. Overall, these results support further studies of topical niacinamide in transplant patients given the high prevalence of polypharmacy, concerns with oral medications, and willingness to try a new topical product if recommended from their health care provider.

Experimental Design

Study Design

Type: Prospective, randomized, controlled trial

Duration: 12 months

Participants: 20 OTRs with history of ≥5 AKs in the past two years and ≥1 prior NMSC Materials: 5% topical niacinamide in a vanicream base will be purchased from The Burgh Pharmacy and provided to participants. No other active ingredients will be added.

Randomization: 1:1 into two arms:

Arm A (Intervention): Topical 5% niacinamide cream applied once daily + SPF 30 sunscreen daily and every 2 hours when outdoors.

Arm B (Control): SPF 30 sunscreen daily and every 2 hours when outdoors. Inclusion Criteria: Age ≥18; History of solid organ transplantation; At least 5 AKs in the past year and prior history of non-melanoma skin cancer Exclusion Criteria: Known allergy to niacinamide or sunscreen components Outcome Measures

Primary Outcome:

Change in AK count at 6 and 12 months, measured by standardized assessment and clinical quantification (see below)

Secondary Outcomes:

Incidence of new keratinocyte carcinomas, confirmed by a board-certified pathologist from histological evaluation Tolerability and adverse events Patient adherence and experience; this will be analyzed using a RedCap survey at the end of the study Quantification: Actinic keratoses and non-melanoma skin cancers will be quantified at regular 6 and 12-month follow-up visits using a standardized scale and transparent sheet for record keeping.

This will be performed using previously published methods by Jansen and Olsen (see below). The severity of each actinic keratosis will be graded with the Olsen scale: 1=mild, 2=moderate or 3=severe. In this classification system, lesions are graded as Olsen Grade I when they are slightly palpable and more easily felt than seen; as Olsen Grade II when the lesions are moderately thick and easy to see and feel; and graded as Olsen Grade III when the lesions are very thick hyperkeratotic AK.

Data Analysis Plan: Comparative analyses of clinical outcomes will be conducted to evaluate the efficacy of the intervention. Differences in actinic keratosis (AK) counts between study arms will be analyzed using two-sample t-tests, and comparisons of incident non-melanoma skin cancer (NMSC) counts will likewise be performed using t-tests, using paired and unpaired approaches. Quantitative findings will be visualized through appropriately scaled bar charts, line graphs, and heat maps to facilitate interpretation of between-group differences. Patient-reported outcomes will include both structured survey responses and open-ended questions. Quantitative survey responses will be analyzed using standard statistical methods, while qualitative responses will undergo systematic content analysis to identify salient themes and patient perspectives.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 History of solid organ transplantation At least 5 AKs in the past year or prior history of skin cancer Participants are willing to continue using SPF30 sunscreen from their own supply

Exclusion Criteria:

Known allergy to niacinamide or sunscreen components Eczema or other skin conditions for which niacinamide is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in baseline AK count | Baseline, 6 months and 12 months
  Change in actinic keratosis count at 6 and 12 months from baseline, measured by standardized assessment and clinical quantification

SECONDARY OUTCOMES:
New NMSC | 6 months and 12 months
  New nonmelanoma skin cancers (NMSC) at 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UPMC Falk Dermatology, Pittsburgh, Pennsylvania
  - UPMC St Margarets Dermatology, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared (age, sex, past medical history, medications, dermatologic history) however this will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: It will be available when the study is complete and for 2 year or longer.
Access Criteria: Those requesting IPD who have a data sharing agreement will be able to access the data. They must request an agreement to the study team.

REFERENCES:
- [Background] Zhang H, George-Washburn EA, Hashemi KB, Cho E, Walker J, Weinstock MA, Bostom A, Robinson-Bostom L, Gohh R. Oral Nicotinamide for Actinic Keratosis Prevention in Kidney Transplant Recipients: A Pilot Double-Blind, Randomized, Placebo-Controlled Trial. Transplant Proc. 2023 Nov;55(9):2079-2084. doi: 10.1016/j.transproceed.2023.06.016. Epub 2023 Oct 12. PMID 37838527
- [Background] Zalaudek I, Piana S, Moscarella E, Longo C, Zendri E, Castagnetti F, Pellacani G, Lallas A, Argenziano G. Morphologic grading and treatment of facial actinic keratosis. Clin Dermatol. 2014 Jan-Feb;32(1):80-7. doi: 10.1016/j.clindermatol.2013.05.028. PMID 24314380
- [Background] Whitley MJ, Suwanpradid J, Lai C, Jiang SW, Cook JL, Zelac DE, Rudolph R, Corcoran DL, Degan S, Spasojevic I, Levinson H, Erdmann D, Reid C, Zhang JY, Robson SC, Healy E, Havran WL, MacLeod AS. ENTPD1 (CD39) Expression Inhibits UVR-Induced DNA Damage Repair through Purinergic Signaling and Is Associated with Metastasis in Human Cutaneous Squamous Cell Carcinoma. J Invest Dermatol. 2021 Oct;141(10):2509-2520. doi: 10.1016/j.jid.2021.02.753. Epub 2021 Apr 20. PMID 33848530
- [Background] Torres-Moral T, Tell-Marti G, Bague J, Roses-Gibert P, Calbet-Llopart N, Mateu J, Perez-Anker J, Potrony M, Alejo B, Iglesias P, Espinosa N, Orte Cano C, Cinotti E, Del Marmol V, Fontaine M, Miyamoto M, Monnier J, Perrot JL, Rubegni P, Tognetti L, Suppa M, Demessant-Flavigny AL, Le Floc'h C, Prieto L, Malvehy J, Puig S. Evaluation of the Biological Effect of a Nicotinamide-Containing Broad-Spectrum Sunscreen on Photodamaged Skin. Dermatol Ther (Heidelb). 2024 Dec;14(12):3321-3336. doi: 10.1007/s13555-024-01298-7. Epub 2024 Nov 7. PMID 39509031
- [Background] Thompson BC, Halliday GM, Damian DL. Nicotinamide enhances repair of arsenic and ultraviolet radiation-induced DNA damage in HaCaT keratinocytes and ex vivo human skin. PLoS One. 2015 Feb 6;10(2):e0117491. doi: 10.1371/journal.pone.0117491. eCollection 2015. PMID 25658450
- [Background] Sivapirabu G, Yiasemides E, Halliday GM, Park J, Damian DL. Topical nicotinamide modulates cellular energy metabolism and provides broad-spectrum protection against ultraviolet radiation-induced immunosuppression in humans. Br J Dermatol. 2009 Dec;161(6):1357-64. doi: 10.1111/j.1365-2133.2009.09244.x. Epub 2009 Apr 20. PMID 19804594
- [Background] Olsen EA, Abernethy ML, Kulp-Shorten C, Callen JP, Glazer SD, Huntley A, McCray M, Monroe AB, Tschen E, Wolf JE Jr. A double-blind, vehicle-controlled study evaluating masoprocol cream in the treatment of actinic keratoses on the head and neck. J Am Acad Dermatol. 1991 May;24(5 Pt 1):738-43. doi: 10.1016/0190-9622(91)70113-g. PMID 1869646
- [Background] Park J, Halliday GM, Surjana D, Damian DL. Nicotinamide prevents ultraviolet radiation-induced cellular energy loss. Photochem Photobiol. 2010 Jul-Aug;86(4):942-8. doi: 10.1111/j.1751-1097.2010.00746.x. Epub 2010 May 13. PMID 20492562
- [Background] Moloney FJ, Comber H, O'Lorcain P, O'Kelly P, Conlon PJ, Murphy GM. A population-based study of skin cancer incidence and prevalence in renal transplant recipients. Br J Dermatol. 2006 Mar;154(3):498-504. doi: 10.1111/j.1365-2133.2005.07021.x. PMID 16445782
- [Background] Martinez JC, Otley CC, Stasko T, Euvrard S, Brown C, Schanbacher CF, Weaver AL; Transplant-Skin Cancer Collaborative. Defining the clinical course of metastatic skin cancer in organ transplant recipients: a multicenter collaborative study. Arch Dermatol. 2003 Mar;139(3):301-6. doi: 10.1001/archderm.139.3.301. PMID 12622621
- [Background] Jansen MHE, Kessels JPHM, Nelemans PJ, Kouloubis N, Arits AHMM, van Pelt HPA, Quaedvlieg PJF, Essers BAB, Steijlen PM, Kelleners-Smeets NWJ, Mosterd K. Randomized Trial of Four Treatment Approaches for Actinic Keratosis. N Engl J Med. 2019 Mar 7;380(10):935-946. doi: 10.1056/NEJMoa1811850. PMID 30855743
- [Background] Hwang JC, Savage KT, Pugliano-Mauro M. Nicotinamide for secondary keratinocyte carcinoma prevention in solid organ transplant recipients. Arch Dermatol Res. 2025 Jun 11;317(1):807. doi: 10.1007/s00403-025-04296-7. PMID 40498148
- [Background] Gensler HL. Prevention of photoimmunosuppression and photocarcinogenesis by topical nicotinamide. Nutr Cancer. 1997;29(2):157-62. doi: 10.1080/01635589709514618. PMID 9427980
- [Background] Damian DL, Patterson CR, Stapelberg M, Park J, Barnetson RS, Halliday GM. UV radiation-induced immunosuppression is greater in men and prevented by topical nicotinamide. J Invest Dermatol. 2008 Feb;128(2):447-54. doi: 10.1038/sj.jid.5701058. Epub 2007 Sep 20. PMID 17882270
- [Background] Chen AC, Martin AJ, Choy B, Fernandez-Penas P, Dalziell RA, McKenzie CA, Scolyer RA, Dhillon HM, Vardy JL, Kricker A, St George G, Chinniah N, Halliday GM, Damian DL. A Phase 3 Randomized Trial of Nicotinamide for Skin-Cancer Chemoprevention. N Engl J Med. 2015 Oct 22;373(17):1618-26. doi: 10.1056/NEJMoa1506197. PMID 26488693
- [Background] Allen NC, Martin AJ, Snaidr VA, Eggins R, Chong AH, Fernandez-Penas P, Gin D, Sidhu S, Paddon VL, Banney LA, Lim A, Upjohn E, Schaider H, Ganhewa AD, Nguyen J, McKenzie CA, Prakash S, McLean C, Lochhead A, Ibbetson J, Dettrick A, Landgren A, Allnutt KJ, Allison C, Davenport RB, Mumford BP, Wong B, Stagg B, Tedman A, Gribbin H, Edwards HA, De Rosa N, Stewart T, Doolan BJ, Kok Y, Simpson K, Low ZM, Kovitwanichkanont T, Scolyer RA, Dhillon HM, Vardy JL, Chadban SJ, Bowen DG, Chen AC, Damian DL. Nicotinamide for Skin-Cancer Chemoprevention in Transplant Recipients. N Engl J Med. 2023 Mar 2;388(9):804-812. doi: 10.1056/NEJMoa2203086. PMID 36856616